CLINICAL TRIAL: NCT05639166
Title: A Phase 2, Randomized, Double-blind, Multicentre, Placebo-controlled Study in Adults to Assess the Safety and Efficacy of Inhaled IBIO123, for Post-exposure Prophylaxis of COVID-19
Brief Title: Study in Adults to Assess the Safety and Efficacy of Inhaled IBIO123, for Post-exposure Prophylaxis of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immune Biosolutions Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IBIO-INH-003
Record Dates: First submitted 2022-12-03; First posted 2022-12-06 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: IBIO; IBIO123; Prophylaxis; Inhalation; monoclonal antibodies; Prevention
MeSH Terms: conditions — COVID-19; Respiratory Aspiration | interventions — IBIO123

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): IBIO123 10 mg
  Interventions: Biological: IBIO123
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IBIO123 — IBIO123 10 mg
  Arms: Active
Other: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, multicentre, placebo-controlled study in adults to assess the safety and efficacy of inhaled IBIO123, for post-exposure prophylaxis of COVID-19.

This study aims to evaluate the efficacy and the safety of IBIO123 and the prophylaxis effect of IBIO123 in participants exposed to COVID-19 in the setting of current and uninterrupted household contacts.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicentre, placebo-controlled study eligible patients will be randomized in a 1:1 ratio to receive either 10mg of IBIO123 or matching vehicle (placebo). IBIO123 will be administered by inhalation via an Aerogen Ultra mesh nebulizer according to the manufacturer's recommendation. Patients will be followed up for a total period of 14 days after the administration of study intervention to detect an infection to SARS-CoV-2.

This study will enroll a total of 140 participants (70 participants on IBIO123 & 70 participants on Placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Are ≥18 years of age at the time of randomization
2. Subject has a household contact with a confirmed COVID-19 cohabiting individual as subject. Initial diagnosis of the COVID-19 positive individual has been within 3 days of screening. COVID-19 positive result (PCR or Antigen) must have been performed by an accredited lab or medical professional. Current and uninterrupted household contacts were defined as family members or close relatives who had unprotected contact with the index case.
3. Subject must have a negative result with the study provided rapid antigen test at baseline and be COVID-19 symptom free.
4. Are men or non-pregnant women. Reproductive and Contraceptive agreements and guidance is provided in Appendix 2. Contraceptive use by men or women should be consistent with local regulations for those participating in clinical studies.
5. Understand and agree to comply with planned study procedures
6. Agree to the collection of nasopharyngeal swabs
7. The participant or legally authorized representative gives signed informed consent as described in Section 10.1.1.2 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. A positive COVID-19 result (PCR or antigen test) within 30 days of screening.
2. Presence of typical COVID-19 symptoms which cannot be explained by another underlying condition (fever >38°C, Oxygen saturation (SpO2) below 93%, dyspnea, difficulty breathing, chills, ageusia, anosmia, cough, myalgia) in the past 48 hours prior to screening.
3. Hypersensitivity to any component of IBIO123
4. Participants who have been previously administered IBIO123.
5. Have received treatment with a SARS-CoV-2 specific monoclonal antibody
6. Have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed.
7. Are pregnant or breast feeding
8. Are investigator site personnel directly affiliated with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Characterize the effect of IBIO123 compared to placebo on laboratory-confirmed COVID-19 infections between baseline and Day 14 | From Baseline to Day 14
  • Proportion of participants who had a laboratory-confirmed COVID-19 infection between baseline and Day 14

SECONDARY OUTCOMES:
Characterize the effect of IBIO123 compared to placebo on laboratory-confirmed COVID-19 infections between baseline and Day 7 | From Baseline to Day 7
  Proportion of participants who had a laboratory-confirmed COVID-19 infection between baseline and Day 7
Characterize the effect of IBIO123 compared to placebo on laboratory-confirmed COVID-19 asymptomatic infections between baseline and Day 7 | From Baseline to Day 7
  Proportion of participants who had a laboratory-confirmed asymptomatic COVID-19 infection between baseline and Day 7
Characterize the effect of IBIO123 compared to placebo on laboratory-confirmed COVID-19 asymptomatic infections between baseline and Day 14 | From Baseline to Day 14
  Proportion of participants who had a laboratory-confirmed asymptomatic COVID-19 infection between baseline and Day 14
Characterize the effect of IBIO123 compared to placebo on overall participant clinical status | From Baseline to Day 14
  Proportion (percentage) of participants who experience these events by Day 14
  * Hospitalisation
  * Mortality
Characterize the effect of IBIO123 compared to placebo on SARS-CoV-2 related symptoms | From Baseline to Day 14
  * Time to symptom onset
  * Proportion of participants demonstrating symptom resolution on Days 7 & 14.
  * Proportion of participants demonstrating Mild, Moderate and Severe symptoms between baseline to Day 7 and day 14
Characterize the effect of IBIO123 compared to placebo on safety and tolerability | From Baseline to Day 14
  Safety assessments such as adverse events (AEs) and Serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Labbe, PhD, Study Director — Immune Biosolutions
Locations (5):
- Jongaie Research, Pretoria West, Pretoria, South Africa
- Ukraine (4):
  - Central City Clinical Hospital of Chernivtsi City Council, Chernivtsi, Chernivetska
  - City Clinical Hospital #1 of Ivano-Frankivsk City Council, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Central C.H. of Ivano-Frankivsk, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Volyn Regional Clinical Hospital, Lutsk, Volyn Oblast